CLINICAL TRIAL: NCT04534127
Title: A Safety and Effectiveness Study of Intratumoral Diffusing Alpha Radiation Emitters for the Treatment of Malignant Cutaneous, Mucosal or Superficial Soft Tissue Neoplasia
Brief Title: Alpha Radiation Emitters Device (DaRT) for the Treatment of Cutaneous, Mucosal or Superficial Soft Tissue Neoplasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-CMN-02_
Record Dates: First submitted 2020-08-18; First posted 2020-09-01 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-11

CONDITIONS: Skin Cancer; Mucosal Neoplasm of Oral Cavity; Soft Tissue Neoplasm
Keywords: Squamous Cell Carcinoma; SCC; Skin Cancer; Skin metastasis; HNSCC; Carcinoma, Squamous; CMN; Basal cell carcinoma; Superficial sarcoma; Kaposi sarcoma; Alpha radiation; Cutaneous lesion; Tongue cancer; Lip cancer; Brachytherapy
MeSH Terms: conditions — Skin Neoplasms; Soft Tissue Neoplasms; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Basal Cell; Sarcoma, Kaposi; Tongue Neoplasms; Lip Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT)

INTERVENTIONS:
Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT) — An intratumoral insertion of a seed(s), loaded with Radium-224, securely fixed in the seeds. The seeds release by recoil into the tumor short-lived alpha-emitting atoms.
  Other Names: DaRT

SUMMARY:
A unique approach for cancer treatment employing intratumoral diffusing alpha radiation emitter device for superficial cutaneous, mucosal or soft tissue neoplasia

DETAILED DESCRIPTION:
This will be a prospective, open label, single arm, controlled study, assessing the safety and efficacy of diffusing alpha emitters radiation therapy (DaRT) delivered through radioactive seeds inserted into the tumor.

This approach combines the advantages of local intratumoral irradiation of the tumor, as used in conventional brachytherapy, with the power of the alpha radiation emitting atoms, that will be introduced in quantities considerably lower than radiation therapy already used in patients.

Superficial lesions with histopathological confirmation of malignancy will be treated using DaRT seeds.

Reduction in tumor size 70 days after DaRT insertion will be assessed. Safety will be assessed by the incidence, severity and frequency of all Adverse Events (AE).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histopathological confirmation of primary or secondary malignant cutaneous neoplastic lesions, or oral cavity mucosal tumors, or superficial soft tissue sarcoma. Confirmation obtained within 6 months of planned treatment.
* Subjects with a tumor size ≤ 7 centimeters in the longest diameter.
* Targetable lesion must be technically amenable for complete coverage (including margins) by the DaRT seeds
* Brachytherapy indication validated by a multidisciplinary team
* Patients who have either failed first-line treatment, or are medically unfit for standard of care (surgery, external-beam radiation therapy or chemotherapy), or refuse standard of care.
* Measurable disease according to RECIST v1.1.
* Subjects over 18 years old.
* Subjects' ECOG Performance Status Scale is < 2.
* Subjects' life expectancy is more than 6 months.
* Platelet count ≥100,000/mm3.
* WBC ≥ 3500/μl, granulocyte ≥ 1500/μl
* AST and ALT ≤ 2.5 X ULN
* International normalized ratio of prothrombin time ≤1.8.
* Creatinine ≤1.9 mg/dL. Women of childbearing potential (WOCBP) will have evidence of negative pregnancy test and are required to use an acceptable contraceptive method to prevent pregnancy for 3 months after brachytherapy.
* Subjects are willing to sign an informed consent form.

Exclusion Criteria:

* Subject has a tumor of Keratoacanthoma histology.
* Known hypersensitivity to any of the components of the treatment.
* Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 12 months.
* Any medical or psychiatric illness which in the opinion of the investigator would compromise the patient's ability to tolerate this treatment or interfere with the study endpoints.
* Patients undergoing systemic immunosuppressive therapy excepting intermittent, brief use of systemic corticosteroids
* Patient requires treatment which may conflict with the endpoints of this study including evaluation of response or toxicity of DaRT
* Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT.
* Patients must agree to use adequate contraception (vasectomy or barrier method of birth control) prior to study entry, for the duration of study participation and for 3 months after discontinuing therapy.
* High probability of protocol non-compliance (in opinion of investigator).
* Subjects not willing to sign an informed consent.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Tumor response to DaRT | 9-11 weeks post DaRT insertion
  Assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1)
Adverse Events | Up to 24 Months
  The incidence, frequency, severity and causality of acute adverse events related to the DaRT treatment according to Common Terminology and Criteria for adverse events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Change in tumor volume | 9-11 weeks post DaRT insertion
  Based on imaging
DaRT seeds placement | 1 Day of procedure
  Assessment by localization of the DaRT seeds in the tumor using CT imaging on the day of DaRT insertion
Change in quality of life | Day 15, Day 30, Day 70, Day 180 post DaRT insertion
  Assessment of patient reported health-related Quality of Life outcome after DaRT, using QoL questionnaire Skindex-16 questionnaire score
Change in quality of life | Day 30, Day 70, Day 180 post DaRT insertion
  Assessment of patient reported health-related Quality of Life outcome after DaRT, using QoL questionnaire Skin Cancer Index (SCI) questionnaire score
Progression Free Survival | 24 months post DaRT insertion
  Time elapsed from response to disease progression

OTHER OUTCOMES:
Adverse Events | Up to 24 Months
  All Adverse Events (AE) related and unrelated to the study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Aron Popovtzer, Principal Investigator — Sharett institute, Hadassah University Hospital - Ein-Kerem
Locations (1):
- Sharett institute, Hadassah Medical Center - Ein-Kerem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No